CLINICAL TRIAL: NCT04993729
Title: A Multicenter, Double-blind, Randomized and Placebo-controlled Pivotal Phase 3 Study to Evaluate the Safety and Efficacy of T89 in the Prevention and Treatment of Acute Mountain Sickness (AMS) After Rapid Ascent
Brief Title: Safety and Efficacy of T89 in the Prevention and Treatment of Adults With Acute Mountain Sickness (AMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T89-31-AMS
Record Dates: First submitted 2021-07-14; First posted 2021-08-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Acute Mountain Sickness (AMS)
Keywords: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- T89 low-dose group (Experimental): Subjects in this group will take three T89 capsules and one Placebo capsule each time by oral administration three times daily for 5 days.
  Interventions: Drug: T89 capsule; Drug: Placebo capsule
- T89 high-dose group (Experimental): Subjects in this group will take four T89 capsules each time by oral administration three times daily for 5 days.
  Interventions: Drug: T89 capsule
- Placebo group (Placebo Comparator): Placebo capsule does not contain any amount of active substance. Subjects in this group will take four placebo capsules each time by oral administration three times daily for 5 days.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: T89 capsule — T89 capsule (trade name Dantonic®) is a botanical drug containing 75mg active substance which is the water extract of Danshen and Sanqi.
  T89 capsules, p.o. TID.
  Arms: T89 high-dose group; T89 low-dose group
Drug: Placebo capsule — Placebo capsules, p.o. TID.
  Arms: Placebo group; T89 low-dose group

SUMMARY:
The specific aim of this double blind, randomized phase III trial is to evaluate the safety and efficacy of T89 in preventing Acute Mountain Sickness (AMS) and relieving the symptoms of AMS after rapid ascent.

DETAILED DESCRIPTION:
Acute mountain sickness (AMS) is a common ailment in people venturing over 2,500 meters altitude. It is a pathological effect of high altitude on humans, caused by acute exposure to low partial pressure of oxygen at high altitude. It presents with a cluster of nonspecific symptoms including headache and one of the following: gastrointestinal symptoms, fatigue and/or weakness, dizziness/ lightheadedness or difficulty sleeping.

T89 capsule is a modernized industrialized version of a traditional Chinese herbal medicine. It is a botanical drug product for oral use. Previous clinical studies showed T89 has substantial benefits in the prevention or amelioration of symptoms associated with acute mountain sickness (AMS).This is double-blind, randomized, placebo controlled pivotal phase 3 study. After informed consent is obtained, eligible subjects will be randomized to one of the 3 study groups (T89 high dose, T89 low dose and placebo control). The study drug will be given orally for 5 days (2 days at sea level and 3 days at high altitude). The clinical assessment of Lake Louise Scoring System (LLSS), blood oxygen saturation, the exercise tolerance, blood pressure and heart rate will be performed at sea level and altitude. A total of 846 subjects will be enrolled with 282 subjects in each treatment arm, and a minimum of 756 subjects are expected to complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers: ages 18 - 55 years old;
2. Primary residence elevation of 2,461 ft (750m) or lower;
3. Not ascending to altitude >10,000 ft within 4 months prior to screening;
4. Females of childbearing potential must have a negative pregnancy test and established on a method of contraception that in the investigator's opinion is acceptable. Females must agree to remain on their established method of contraception from the time of the screening visit and throughout the study period;
5. Willing to participate voluntarily and sign a written informed consent.

Exclusion Criteria:

1. Subjects with medical history of cardiovascular, cerebrovascular diseases or asthma; uncontrolled hypertension with SBP>140 and or DBP>90 mmHg;
2. Subjects with current and clinically significant respiratory system disease, digestive disease, liver disease, central nervous system disease, psychiatric disease, metabolic disease, renal disease, acute infection or anemia, or who test positive for COVID-19 (COVID testing will be performed, not per study requirement, but in compliance with local law or policy, and subject with known positive for COVID-19 will be excluded).
3. Total LLSS score (LLSS score) is ≥2 at any check point during screening period;
4. Blood oxygen saturation (SpO2), preferably tested on the left-hand index finger, is less than 95% at screening visits;
5. Subjects with abnormal renal or liver function with clinical significance (ALT or AST > 2×ULN, Creatinine > ULN) at screening visit;
6. Subjects with CRP > ULN at screening visit;
7. Subjects with primary (migraine, tension-type headache, and cluster headache etc.) or secondary headaches (headache related to infection, vascular disease etc.) within one month at screening;
8. Surgery or blood donation within 3 months prior to screening;
9. On treatment of any medications (including any dietary supplements) except for birth control within 14 days prior to screening and throughout the study period;
10. Smokers who had a habit of smoking during the last 4 months prior to the starting of screening;
11. Contradictive to treatment of Danshen (Radix Saliva Miltiorrhize Bge., RSM) products;
12. Women who are pregnant or lactating.
13. Substance abuse. Subjects with a recent (within the last 6 months) history of substance abuse (alcohol, marijuana, or known drug dependence). Or subjects who have a positive urine substance test at screening;
14. Participation in any other interventional clinical trial or on an investigational drug within 30 days prior to screening;
15. A family member or relative of the study site staff;
16. Any condition that, in the opinion of the investigator, is likely to prevent compliance with the study protocol, interfere with the assessment, or pose a safety concern if the subject participates in the study at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 853 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Change of baseline corrected mean LLSS score on Day 4 morning (next mornings after arrival at high altitude) between T89 and placebo groups. | Baseline and day 4
  2018 Lake Louise Scoring System (LLSS) score [0-12] will be used in this primary outcome assessment. The higher LLSS scores mean the worse symptoms of AMS. Baseline will be the average of LLSS scores on Day 2 and the one on Day 3 before breakfast.

SECONDARY OUTCOMES:
The change of blood oxygen saturation levels (SpO2) at high altitude between T89 and placebo groups. | Baseline and days 3-6
  Blood oxygen saturation (SpO2) will be measured by pulse oximeter at sea level (on screening day, Day 2 and Day 3 morning) and at high altitude (Day 3 after arriving and Day 4-Day 6).
The change of the area under the curve (AUC) of baseline corrected LLSS score-time profile between T89 and placebo groups. | Baseline and days 3-6
  AUC of based corrected LLSS score-time curve during altitude stay will be compared between T89 and placebo groups.
The change in total incidence of LLSS score ≥5 on Day 4 morning between T89 and placebo groups. | Day 4 morning
  Total incidence of LLSS score ≥5 will be recorded on Day 4 morning. The difference between T89 and placebo groups will be compared.
The change of percentage reduction of the daily total LLSS score from Day 4 to Day 5 between T89 and placebo groups. | Days 4-5
  Proportional reduction of the daily total LLSS score from Day 4 to Day 5 at high altitude will be compared between T89 and placebo groups.
The change of baseline corrected LLSS score at any given time points between T89 and placebo groups. | Baseline and days 3-6
  2018 Lake Louise Scoring System (LLSS) score [0-12] will be used in this primary outcome assessment. The higher LLSS scores mean the worse symptoms of AMS. Baseline corrected LLSS score will be assessed at every time points at high altitude from Day 3 to Day 6.
The change of total functional LLSS score at any given time points between T89 and placebo groups. | Baseline and days 3-6
  The functional score [0-3] will be self-reported using the 1993 Lake Louise Acute Mountain Sickness Score System to evaluate how did AMS symptoms affect subjects' activities, if they have AMS symptoms. The higher functional scores mean the worse symptoms of AMS.
Accumulated incidence rate of subjects who underwent any rescue activity in transit and after ascending between T89 and placebo groups. | Days 3-6
  The total incidence of subjects who received rescue medicine, oxygen or descent to lower level will be recorded in transit and after arriving high altitude.
The change of exercise tolerance at high altitude (on Day 3 after arriving and Day 5, respectively) from those of at sea level baseline between T89 and placebo groups. | Baseline and days 3 and 5
  Exercise tolerance test will be performed on bicycle ergometer.
The change of the symptom-related AE drop-out rate between T89 and placebo groups. | Days 3-6
  The symptom-related AE drop-out rate is proportion of participants who dropped out study because of adverse event.
The change of blood pressure (mmHg) during at high altitude from those of at sea level baseline on Day 1 (prior to the first dose administration) between T89 and placebo groups. | Screening day, days 2-6
  Unit of blood pressure is mmHg. Both systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be recorded. Blood pressure will be measured at each applicable visit during the whole study period (screening day, Day 2-Day 6).
The change of heart rate (beats/minute) at high altitude from those of at sea level baseline on Day 1 (prior to the first dose administration) between T89 and placebo groups. | Screening day, days 2-6
  Unit of heart rate is beats/minute. Heart rate will be measured at each applicable visit during the whole study period (screening day, Day 2-Day 6).

CONTACTS AND LOCATIONS:
Overall Officials: Henry H Sun, PhD, MD, Study Chair — Tasly Pharmaceuticals, Inc.
Locations (3):
- Hypoxia Research Lab, UCSF Parnassus Campus, S-256, San Francisco, California, United States
- China (2):
  - Affiliated Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Tibet Autonomous Region People's Hospital, Lhasa, Tibet

IPD SHARING:
Plan to Share IPD: No